CLINICAL TRIAL: NCT02643680
Title: Clinical Efficacy of the Novel Biocellulose Wound Dressing Containing Silk Sericin and Polyhexamethylene Biguanide for Split-thickness Skin Graft Donor Sites
Brief Title: Clinical Study of Biocellulose Wound Dressing Containing Silk Sericin and PHMB for STSG Donor Sites
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Med CU IRB 242/58
Record Dates: First submitted 2015-12-16; First posted 2015-12-31 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Wound; Disorder of Skin Donor Site
Keywords: Biocellulose; Silk sericin; Polyhexamethylene biguanide; Split thickness skin graft donor site
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The novel biocellulose wound dressing (Experimental)
  Interventions: Device: The novel biocellulose wound dressing
- Bactigras (Active Comparator)
  Interventions: Device: Bactigras

INTERVENTIONS:
Device: The novel biocellulose wound dressing — The novel biocellulose dressing will used as a primary dressing at one half of the donor site. Then,the wound will be covered with 2 layers of gauze (secondary dressing) and 1 layer of bandage.The primary dressing will be unchanged until the wound healing (the day that the dressing detaches by itself with no exudate and air contacted pain) except signs of infection. The secondary dressing will be changed when excessive fluid appears.
  Other Names: Biocellulose dressing containing silk sericin and PHMB
  Arms: The novel biocellulose wound dressing
Device: Bactigras — Bactigras will used as a primary dressing at another one half of the donor site. Then,the wound will be covered with 2 layers of gauze (secondary dressing) and 1 layer of bandage.The primary dressing will be unchanged until the wound healing (the day that the dressing detaches by itself with no exudate and air contacted pain) except signs of infection. The secondary dressing will be changed when excessive fluid appears.
  Other Names: Chlorhexidine acetate 0.5% in white soft paraffin
  Arms: Bactigras

SUMMARY:
1. The wound healing time of STSG donor sites which are treated with the novel biocellulose wound dressing containing silk sericin and PHMB should be less or equal to Bactigras®.
2. The wound quality of STSG donor sites which are treated with the novel biocellulose wound dressing containing silk sericin and PHMB should be less or equal to Bactigras®.
3. The amounts of STSG donor site infection which are treated with the novel biocellulose wound dressing containing silk sericin and PHMB should not be more than Bactigras®.
4. The pain level of STSG donor sites which are treated with the novel biocellulose wound dressing containing silk sericin and PHMB should be less or equal to Bactigras®.
5. Adverse events which are occurred from the novel biocellulose wound dressing containing silk sericin and PHMB treatment for STSG donor sites and Bactigras® will be reported, if they occur.

DETAILED DESCRIPTION:
The goals of STSG donor site treatment are to accelerate wound healing, prevent infection, reduce pain, and maintain an optimal environment healing promotion. Biocellulose is an ultrafine fiber structure that can hold a large amount of water and has a cooling effect that decreases pain without causing an allergic reaction or irritation.Silk sericin (SS) can activate the growth of fibroblast cells which promote collagen type I production and accelerated wound healing without toxicity . Polyhexamethylene biguanide (PHMB) is a broad spectrum antimicrobial agent with high efficacy and low toxicity. Therefore, the combination of silk sericin and PHMB in biocellulose dressings would benefit STSG donor site wound treatment. The purpose of this study is to investigate the clinical efficacy of this dressing for STSG donor site wound treatment compared with Bactigras® (chlorhexidine acetate 0.5% in white soft paraffin), which is the standard dressing for this type of wound at King Chulalongkorn Memorial Hospital, by monitoring the time required for complete re-epithelization, wound quality, the rate of infection, pain, and the adverse events from December 2015 to November 2016. Thirty two subjects (more than 18 years) with STSG donor site at thigh will be recruited in this study. Block randomization will be used for separation half of eligible wound to cover with novel biocellulose wound dressing containing silk sericin and PHMB or Bactigras®. Wound healing time is the day that the dressing detaches by itself with no exudate and air contacted pain. Wound quality at 1,3,and 6 months will be measured in terms of erythema level, melanin level, transepidermal water loss by using Cutometer® and scar quality (vancouver scar scale). Sign of infection, pain (VAS score), hepatic and renal function will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have STSG donor site wounds on the thigh
* Age more than 18 years old
* Signed consent form

Exclusion Criteria:

* Systemic infection
* Known allergy or hypersensitivity reaction to silk sericin , PHMB, or chlorhexidine acetate
* Known skin diseases
* Known immunocompromised diseases
* Known mental defect or schizophrenia
* Pregnancy or lactation
* Not follow all procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Healing time | 6 months
  The day that the dressing detaches by itself with no exudate and air contacted pain

SECONDARY OUTCOMES:
Erythema and melanin level of wound | 1 year
  Erythema and melanin level by using Cutometer® with mexameter mode (Courage+Khazaka electronic GmbH, Germany) at healing day, 1, 3,and 6 months after healing
Transepidermal water loss of wound | 1 year
  Transepidermal water loss by using Cutometer® with tewameter mode (Courage+Khazaka electronic GmbH, Germany) at healing day, 1, 3,and 6 months after healing
Wound scar formation | 1 year
  Vancouver scar scale at healing day, 1, 3,and 6 months after healing
Signs of infection | 1 year
  Signs of infection: swelling, redness, bad odor, purulent discharge everyday
Swab test of infection wound | 1 year
  Swab evaluation when signs of infection observes
Pain score | 6 months
  Visual analogue scale
Adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pornanong Aramwit, Ph.D, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn Hospital, Bangkok, Thailand